CLINICAL TRIAL: NCT04905771
Title: Characterizing Follicles From Auto-transplanted Ovarian Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter Humaidan (Other)
Collaborators: Reproduktionsbiologisk Laboratorium, JMC, Rigshospitalet, København (Unknown)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: OTT-study2021
Record Dates: First submitted 2021-05-21; First posted 2021-05-28 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Infertility, Female
Keywords: Infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the project is to characterize the hormonal conditions in egg follicles in women who, prior to fertility treatment, have had autotransplanted frozen ovarian tissue for the purpose of fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Has had frozen and later autotransplanted ovarian tissue for fertility preservation purposes
* Included in fertility treatment with eff retrieval at the Fertility Clinic Regional Hospital Skive
* Is willing and able to give informed consent

Exclusion Criteria:

- Patients undergoing fertility treatment but have not received autotransplanted ovarian tissue for fertility preservation purposes

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 30 women undergoing fertility treatment who has had frozen and later autotransplanted ovarian tissue for fertility preservation purposes
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Characterize hormone production in follicles from autotransplanted ovarian tissue | 5 years
  Women undergoing fertility treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Skive Regional Hospital, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No